CLINICAL TRIAL: NCT00435162
Title: A Randomized, Multicenter, Double-blind, 6 Week Study to Evaluate the Dose Response of Valsartan on Blood Pressure Reduction in Children 6 Months - 5 Years Old With Hypertension, Followed by a 2 Week Placebo Withdrawal Period.
Brief Title: Dose Response of Valsartan on Sitting Systolic Blood Pressure in Children 6 Months - 5 Years of Age With High Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAL489K2303
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: Children; pediatrics; High Blood Pressure; Hypertension; Valsartan
MeSH Terms: conditions — Hypertension | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Low Dose (Experimental)
  Interventions: Drug: Valsartan 0.25 mg/kg
- Medium Dose (Experimental)
  Interventions: Drug: Valsartan 1.0 mg/kg
- High Dose (Experimental)
  Interventions: Drug: Valsartan 4.0 mg/kg

INTERVENTIONS:
Drug: Valsartan 0.25 mg/kg — once daily
  Arms: Low Dose
Drug: Valsartan 1.0 mg/kg — once daily
  Arms: Medium Dose
Drug: Valsartan 4.0 mg/kg — once daily
  Arms: High Dose

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of three doses of valsartan (0.25, 1.0, and 4.0 mg/kg) on mean sitting systolic blood pressure (MSSBP) and mean sitting diastolic blood pressure (MSDBP) in 6 months - 5 year old children with hypertension (sitting systolic blood pressure [SSBP] ≥ 95th percentile ).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months - 5 years at Visit 1, with a documented history of hypertension
* Must be able to swallow liquid formulation
* Must be ≥ 6 kg or ≤ 40 kg at randomization
* Must have documented history MSSBP (mean of 3 measurements) must be ≥ 95th percentile for age, gender and height, at randomization
* If patients enter with uncontrolled BP they can remain on background antihypertensives with an unchanged dosing regimen
* If patients have had a solid organ transplant more than 1 year ago they must be on stable doses of immunosuppressive therapy
* Parent(s)/guardian(s) are able to follow verbal and/or written instructions in the local language

Exclusion Criteria:

* Patients with background ARB therapy
* Patients demonstrating any clinically significant abnormalities or clinically noteworthy abnormal lab values (other than those relating to renal function)
* AST/SGOT or ALT/SGPT > 3 times the upper limit of the reference range
* Glomerular filtration rate < 30 mL/min/1.73m²
* Serum potassium > upper limit of the reference range
* MSSBP ≥ 25% above the 95th percentile
* Patients exhibiting clinically significant ECG abnormalities
* Patients that have coarctation of the aorta with a gradient of ≥ 30 mm Hg, or renal artery stenosis

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2007-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Sponsor GmbH
Locations (11):
- Sites in USA, USA, New Jersey, United States
- Sites in Belgium, Belgium, Belgium
- Sites in Brazil, Brazil, Brazil
- Sites in France, Paris, France
- Sites in Hungary, Hungary, Hungary
- Sites in India, India, India
- sites in Italy, Italy, Italy
- Sites in Poland, Poland, Poland
- Sites in South Africa, South Africa, South Africa
- Sites in Sweden, Sweden, Sweden
- Sites in Turkey, Turkey, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At period 1, participants were randomized (2:1:2) to Valsartan 0.25 mg/kg, 1.0 mg/kg or 4.0 mg/kg. At period 2, participants were randomized (1:1) to either stay on Valsartan or switch to placebo.
Groups:
- Low Dose in Both Periods: Valsartan 0.25 mg/kg in both periods
- Low Dose, Then Placebo: Valsartan 0.25 mg/kg, then placebo
- Medium Dose in Both Periods: Valsartan 1.0 mg/kg in both periods
- Medium Dose, Then Placebo; High Dose in Both Periods: Valsartan 1.0 mg/kg, then placebo
- High Dose, Then Placebo: Valsartan 4.0 mg/kg, then placebo
Period: Period 1 (6 Weeks)
Arm/Group | Low Dose in Both Periods | Low Dose, Then Placebo | Medium Dose in Both Periods | Medium Dose, Then Placebo | High Dose in Both Periods | High Dose, Then Placebo
Started | 15 | 15 | 6 | 8 | 15 | 15
Completed | 15 | 15 | 6 | 8 | 15 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (2 Weeks)
Arm/Group | Low Dose in Both Periods | Low Dose, Then Placebo | Medium Dose in Both Periods | Medium Dose, Then Placebo | High Dose in Both Periods | High Dose, Then Placebo
Started | 15 | 15 | 6 | 8 | 15 | 15
Completed | 15 | 14 | 6 | 8 | 15 | 15
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose: Extemporaneous suspension of valsartan 0.25 mg/kg, taken once daily
- Medium Dose: Extemporaneous suspension of valsartan 1.0 mg/kg, taken once daily
- High Dose: Extemporaneous suspension of valsartan 4.0 mg/kg, taken once daily
- Total: Total of all reporting groups
Arm/Group | Low Dose | Medium Dose | High Dose | Total
Number analyzed (Participants) | 30 | 14 | 30 | 74
Age Continuous [Mean (Standard Deviation); unit: years] | 3.4 (1.28) | 3.2 (1.48) | 3.3 (1.53) | 3.3 (1.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 4 | 9 | 26
  Male | 17 | 10 | 21 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure (MSSBP) From Baseline to End of Period 1 (Week 6)
Time Frame: baseline and week 6
Population: Analysis: Intention to Treat Imputation Technique: Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 30 | 14 | 30
mm Hg | -8.3 (10.44) | -10.3 (9.83) | -14.4 (10.93)
Statistical Analysis 1: Comparison: Low Dose vs Medium Dose vs High Dose; Slope change across all 3 active treatment groups; Test type: Superiority or Other; p = 0.0990, Regression, Linear; Slope = -1.05, 95% CI 2-sided [-2.31 to 0.20]

2. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSDBP)to End of Period 1 (Week 6)
Time Frame: baseline and week 6
Population: Analysis: Intention to Treat Imputation Technique: Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 30 | 14 | 30
mm Hg | -4.7 (9.53) | -8.6 (12.43) | -6.7 (10.61)

3. Secondary Outcome: Change From End of Period 1 (Week 6) in Mean Sitting Systolic Blood Pressure (MSSBP) to End of Placebo-controlled Withdrawal Period (Week 8)
Time Frame: week 6 and week 8
Population: Analysis: Intention to Treat Imputation Technique: Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Valsartan: pooled across all dosage levels
Arm/Group | Valsartan | Placebo
Number analyzed (Participants) | 35 | 38
mm Hg | 2.6 (8.38) | 4.1 (9.66)

4. Secondary Outcome: Change From End of Period 1 (Week 6) in Mean Sitting Diastolic Blood Pressure (MSDBP) to End of Placebo-controlled Withdrawal Period (Week 8)
Time Frame: week 6 and week 8
Population: Analysis: Intention to Treat Imputation Technique: Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan | Placebo
Number analyzed (Participants) | 35 | 38
mm Hg | 1.8 (8.99) | 3.4 (8.74)

ADVERSE EVENTS:
Time Frame: Period 1 (Baseline to Week 6) and Period 2 (Week 6 to Week 8)
Groups:
- High Dose in Both Periods: Valsartan 4.0 mg/kg in both periods
Arm/Group | Low Dose in Both Periods | Low Dose, Then Placebo | Medium Dose in Both Periods | Medium Dose, Then Placebo | High Dose in Both Periods | High Dose, Then Placebo
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 0/6 | 1/8 | 0/15 | 2/15
Other Adverse Events (participants affected / at risk) | 8/15 | 10/15 | 3/6 | 4/8 | 9/15 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose in Both Periods (N=15) | Low Dose, Then Placebo (N=15) | Medium Dose in Both Periods (N=6) | Medium Dose, Then Placebo (N=8) | High Dose in Both Periods (N=15) | High Dose, Then Placebo (N=15)
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose in Both Periods (N=15) | Low Dose, Then Placebo (N=15) | Medium Dose in Both Periods (N=6) | Medium Dose, Then Placebo (N=8) | High Dose in Both Periods (N=15) | High Dose, Then Placebo (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 2 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2 | 3
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Scarlet fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.